CLINICAL TRIAL: NCT02054039
Title: Comparison Between Incentive Spirometry and Breath Stacking After Cardiac Surgery
Brief Title: Incentive Spirometry and Breath Stacking
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Eliane Regina Ferreira Sernache de Freitas, Eliane Regina Ferreira Sernache de Freitas, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 186.780
Record Dates: First submitted 2014-02-01; First posted 2014-02-04 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Complications
Keywords: Cardiac surgery; Spirometry; Physical Therapy Modalities; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incentive spirometry (IS) (Experimental): Group I
  Interventions: Device: Incentive spirometry (IS)
- Breath stacking (BS) (Active Comparator): Group II
  Interventions: Device: Breath Stacking (BS)

INTERVENTIONS:
Device: Incentive spirometry (IS) — Mechanical devices activated by an inspiratory effort, which is viewed by the elevation of a plateau or balls in a transparent cylinder having a calibrated scale that displays the inspired flow.
  Arms: Incentive spirometry (IS)
Device: Breath Stacking (BS) — Equipment with a one-way valve that masks and promotes the accumulation of successive inspiratory volumes, preventing expiration
  Arms: Breath stacking (BS)

SUMMARY:
- Postoperative pulmonary complications in patients undergoing cardiac surgery are a major clinical problem, presenting negative impact on morbidity, mortality , length of hospital stay and health care costs. Although physical therapy has been widely used as a resource to improve lung function in the postoperative period, the adoption of routine procedures of physical therapy needs be discussed.

* Incentive spirometers are mechanical devices used to reduce postoperative pulmonary complications. In general, they are activated by an inspiratory effort, visualized by an uplifted plate or ball in a transparent cylinder during sustained inspiration.
* Breath Stacking is a technique allowing the patient inhale a greater volume of air, kept for a longer period of time using a one-way valve, thus promoting the accumulation of successive inspiratory volume and preventing exhalation.
* The objective of the study is to evaluate the effectiveness of two different techniques of respiratory therapy on both reducing postoperative pulmonary complications and improving lung function.
* Type of study : randomized clinical trial
* Hypothesis

  1. Both techniques Trifllo II Incentive Spirometry ( IS) (Trifllo ® - II ) and Breath Stacking ( BS ) may present similar effectiveness on reducing pulmonary complications, improving lung function and respiratory muscle strength ( MIP and MEP), as well as reducing hospital stay .
  2. Trifllo II Incentive Spirometry ( IS) (Trifllo ® - II ) may be more effective than Breath Stacking on reducing pulmonary complications, improving lung function and respiratory muscle strength, as well as reducing hospital stay.

DETAILED DESCRIPTION:
* Type of study : randomized clinical trial
* Study site: The study will be carried out at the Hospital Santa Casa de Londrina.
* Subjects: all patients scheduled for cardiac surgery will be studied ( CABG and / or valve replacement )
* Patients will be evaluated both preoperatively, and on the fifth postoperative day (POD). They will be informed about the procedures to which they will be submitted, as well as the objective of the proposed study preoperatively. If approved by the patient, the "Statement of Informed Consent - SIC" will be signed.
* Inclusion Criteria

  a. Individuals admitted to the Hospital Santa Casa de Londrina (HSCL) with programming for cardiac surgery with cardiopulmonary bypass, age above 18 years; and referral for surgery by the study teams. Individuals must be aware, informed, and agreed to participate in the study, including signing of SIC.
* Exclusion Criteria a. Individuals with cognitive impairment that prevents the implementation of spirometry (lung function ), manovacuometry (MIP and MEP) and incentive spirometry, below 18 years of age, patients with chronic obstructive pulmonary disease diagnosed by clinical history and spirometry ( FVC < 80 % predicted and / or FEV1 < 70 % predicted ) and individuals with a history of asthma.

b . Patients will be withdrawn from the study and the Intention to Treat Analysis will be performed in the case of: patients who cannot be extubated because of the need for continuing mechanical ventilation after 24 hours of post-operative complications in the postoperative period; hemodynamic instability ; myocardial infarction during operation ; severe blood loss defined by the medical staff; loss of 20 % or more of total blood volume ( 12 ); mean arterial pressure (MAP ) < 70 mmHg,; reduced cardiac output requiring the use of intra-aortic balloon or vasoactive drugs for more than 72 hours, after ICU admission or need for new reintubation. Patients who did not agree to participate by not signing the SIC.

* Procedures and interventions a. randomization

  a.1 . After being selected by the inclusion criteria and had signed the informed consent preoperatively, patients will be allocated to one of two groups based on Consort ;

  a.2 . The allocation will be generated through a standardized random table. The allocation concealment will be ensured using opaque envelopes, sealed, and numbered serially. The envelope containing a card with the treatment will be opened by a secretary responsible for that.
* Formation of groups a. EI Group I - Intervention with flow-oriented incentive spirometry (IS) ( Trifllo ® - II ).

b . BS Group II - Intervention with Breath- Stacking technique (BS).

* Recording and evaluation of the patient: patients included in the study will be recorded and evaluated by a physical therapist involved in the trial (blind) according to the standardized forms.
* Duration of the intervention: Both therapy modalities (Group I and Group II) will be held twice daily during the ICU stay, and once a day during hospitalization in the ward, until the fifth postoperative day. Each session will consist of three sets of five maneuvers.

ELIGIBILITY:
Inclusion Criteria:

• Subjects admitted to the Hospital Santa Casa de Londrina (HSCL) with programming for cardiac surgery with cardiopulmonary bypass, age above 18 years, and referral for surgery by the study teams. Individuals must be aware, informed, and agreed to participate in the study, including signing of SIC

Exclusion Criteria:

* Individuals with cognitive impairment that prevents the implementation of spirometry (lung function ), manovacuometry (MIP and MEP) and incentive spirometry; below 18 years of age; patients with chronic obstructive pulmonary disease diagnosed by clinical history and spirometry ( FVC < 80 % of predicted and / or FEV1 < 70 % predicted); and individuals with a history of asthma.
* Patients will be withdrawn from the study and the Intention to Treat Analysis will be performed in the case of: patients who cannot be extubated because of the need for continuing mechanical ventilation after 24 hours of post-operative complications in the postoperative period; hemodynamic instability ; myocardial infarction during operation ; severe blood loss defined by the medical staff; loss of 20 % or more of total blood volume; mean arterial pressure (MAP ) < 70 mmHg; reduced cardiac output requiring the use of intra-aortic balloon or vasoactive drugs for more than 72 hours, after ICU admission or need for new reintubation. Patients who did not agree to participate by not signing the SIC

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary complications | 18 months
  * Pneumonia
  * Atelectasis
  * Acute respiratory infection

SECONDARY OUTCOMES:
Lung Function | 18 months
  Lung function will be assessed by spirometry, aimed at measuring the forced vital capacity (FVC), forced expiratory volume in one second (VFE1), and the ratio CVF/VFE1
Respiratory muscle strength | 18 months
  Respiratory muscle strength will be assessed by measuring both the maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP). The values obtained for each volunteer on the respective predicted values for the Brazilian population, according to the prediction equations proposed by Neder et al will be compared.

OTHER OUTCOMES:
hospital stay | 18 months
  Length of hospital stay in days, in the immediate postoperative period ( POI ) with the arrival of the patient in the ICU until discharge or death .
Mortality from pulmonary cause | 18 months
  Mortality from pulmonary causes will be derived from primary and secondary causes, and will be considered a medical inference.

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Freitas, PhD, Principal Investigator — Federal University of São Paulo and University of Northern Parana
Locations (1):
- Hospital Santa Casa de Londrina, Londrina, Paraná, Brazil